CLINICAL TRIAL: NCT03782298
Title: Safety and Performance of PEEK Anchors (DYNOMITE, SPYROMITE, RAPTOMITE, FOOTPRINT Ultra PK SL) in Extremities
Brief Title: Safety and Performance of PEEK Anchors in Extremities
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018.15.SMD.PEEK.RET.EXT
Record Dates: First submitted 2018-11-06; First posted 2018-12-20 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2021-11

CONDITIONS: Medial or Lateral Instability Repairs/Reconstructions; Hallux Valgus Repairs; Achilles Tendon Repairs/Reconstructions; Midfoot Reconstructions; Metatarsal Ligament/Tendon Repairs/Reconstructions; Bunionectomy; Scapholunate Ligament Reconstructions; Ulnar; Lateral Epicondylitis Repair; Bicep Tendon Reattachments
Keywords: Dynomite; Spyromite; Raptormite; Foot; Ankle; Wrist; Hand; Elbow; Footprint

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Spyromite, Dynomite, Raptomite, Footprint Ultra PK SL — PEEK Suture Anchors, which include:
  * SPYROMITE™ 2.0 PK Suture Anchor with Needles
  * DYNOMITE™ 2.0 PK Suture Anchor with Needles
  * RAPTORMITE™ 3.0 Suture Anchor with Needles
  * FOOTPRINT™ Ultra PK SL Suture Anchor

SUMMARY:
Safety and performance of the study devices in extremities up to 12 months post-surgery

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have undergone extremity joint repair using the study devices.
* Subjects aged 18 years and older at the time of surgery.

Exclusion Criteria:

* Subject is entered in another investigational drug, biologic, or device study or has been treated with an investigational product within 12 months post-operative.
* Subjects who are < 3 months post-operative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have undergone extremity joint repair using the study devices, PEEK Anchors (DYNOMITE, SPYROMITE, RAPTOMITE, FOOTPRINT Ultra PK SL)
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judth Horner, Study Chair — Smith & Nephew, Inc.
Locations (4):
- United States (3):
  - OrthoCarolina, Charlotte, North Carolina
  - Precision Orthopaedic Specialties, Inc., Chardon, Ohio
  - Foot and Ankle Associates of North Texas-Grapevine, Grapevine, Texas
- Fowler Kennedy Sport Medicine Clinic, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: It was intended to enroll participants for 4 PEEK suture anchor devices; however, no participants were enrolled in the SPYROMITE™ 2.0 PK Suture Anchor with Needles group, resulting in 3 suture anchor groups being analyzed. A total of 140 participants were enrolled in the study and 142 joints were observed. Multiple devices were implanted in 2 participants. Separate "arms" not created as participants had the same procedure on the same joint. Anchors are shown by categories (rows) throughout.
Units Other Than Participants: joints
Groups:
- Polyetheretherketone (PEEK) Extremity Suture Anchors: Participants who have received Polyetheretherketone (PEEK) Extremity Suture Anchors, which included:
  DYNOMITE™ 2.0 PK Suture Anchor with Needles, RAPTORMITE™ 3.0 Suture Anchor with Needles, FOOTPRINT™ Ultra PK SL Suture Anchor
Period: Overall Study
Arm/Group | Polyetheretherketone (PEEK) Extremity Suture Anchors
Started | 140; 142 joints
DYNOMITE™ 2.0 PK Suture Anchor With Needles (Type of suture anchor received at start) | 17; 17 joints
RAPTORMITE™ 3.0 Suture Anchor With Needles (Type of suture anchor received at start) | 71; 71 joints
FOOTPRINT™ Ultra PK SL Suture Anchor (Type of suture anchor received at start) | 57; 59 joints
Completed | 136; 136 joints
Not Completed | 4; 6 joints
Not completed — Protocol Deviation | 4

BASELINE CHARACTERISTICS:
Population: Participants enrolled in the study who had previously undergone extremity repair using PEEK suture anchors (i.e., retrospective data). The type(s) of PEEK anchor used during surgery was surgeon decision on a case by case basis. Multiple anchor types could be used in one surgery if required. 2 participants had multiple devices implanted. Participants with bilateral surgeries had both surgeries recorded independently. Device data analyzed individually dependent on unique suture anchor implanted.
Units Other Than Participants: joints
Arm/Group | Polyetheretherketone (PEEK) Extremity Suture Anchors
Number analyzed (Participants) | 140
Number analyzed (joints) | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (13.6)
Sex: Female, Male [Count of Units; unit: joints]
  Female | 83
  Male | 59
Ethnicity (NIH/OMB) [Count of Units; unit: joints]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 115
  Unknown or Not Reported | 21
Race/Ethnicity, Customized [Count of Units; unit: joints]
  American Indian or Alaska Native: No | 142
  American Indian or Alaska Native: Yes | 0
  Asian: No | 142
  Asian: Yes | 0
  Black or African American: No | 137
  Black or African American: Yes | 5
  Native Hawaiian or Other Pacific Islander: No | 142
  Native Hawaiian or Other Pacific Islander: Yes | 0
  White: No | 22
  White: Yes | 120
  Other: No | 124
  Other: Yes | 18
Location of Device Implantation [Count of Units; unit: joints] — Location of device implantation indicated as left, right, or bilaterally (i.e., both left & right).
  joints
    Left | 72
    Right | 66
    Bilaterally | 4
Duration of Surgery (min) [Mean (Standard Deviation); unit: minutes] — Population: Data only available for 102 participants due to the retrospective nature of the study.
  minutes
    number analyzed (Participants) | 102
    (all) | 67 (28.5)
Duration of time from injury to surgery (days) [Mean (Standard Deviation); unit: days] — Population: Data only available for 87 participants due to the retrospective nature of the study.
  days
    number analyzed (Participants) | 87
    (all) | 508.4 (994.7)
Number of Joints Treated by Indication [Count of Units; unit: joints]
  Medial instability | 58
  Achilles tendon | 54
  Midfoot | 2
  Metatarsal ligament | 11
  Other | 6
  Medial instability & Achilles tendon | 1
  Medial instability & Other | 5
  Midfoot & Metatarsal ligament | 4
  Metatarsal ligament & Other | 1
Disposition of Suture Anchors [Count of Participants; unit: Participants] — Count of participants by unique PEEK Suture Anchors implanted. Population: Information provided based on the unique device implanted. Out of 140 overall participants, 2 were implanted with multiple Suture Anchors (devices).
  Participants
    DYNOMITE™ 2.0 PK Suture Anchor with Needles | 17
    RAPTORMITE™ 3.0 PK Suture Anchor with Needles | 71
    FOOTPRINT™ Ultra PK SL Suture Anchor | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Success of the Study Devices in the Extremity Over a Time Period of 6 Months After Intervention
Description: Clinical success was defined as extremity repairs without signs of device failure and/or re-intervention as assessed by the surgeon. Specifically, clinical success was considered "Yes" based on the following 3 main criteria:
  * no inflammatory or allergic response
  * no device-related adverse event (AE)
  * no device deficiencies (DDs) leading to revision surgery (re intervention) on the index extremity
Time Frame: 6 months
Population: Participants analyzed at time frame specified for each row indicates participant provided retrospective data. Some participants implanted with multiple Suture Anchors (devices). Data analyzed independently based on specific device implanted (i.e., participants with multiple devices analyzed by unique suture anchor). Anchors shown by rows/categories as the same procedure occurred on the same joint. Overall number of participants analyzed shows combined total of distinct participants assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Polyetheretherketone (PEEK) Extremity Suture Anchors
Number analyzed (Participants) | 140
Participants
  DYNOMITE™ 2.0 PK Suture Anchor with Needles: number analyzed (Participants) | 17
  DYNOMITE™ 2.0 PK Suture Anchor with Needles: Yes | 16
  DYNOMITE™ 2.0 PK Suture Anchor with Needles: No | 1
  RAPTORMITE™ 3.0 PK Suture Anchor with Needles: number analyzed (Participants) | 71
  RAPTORMITE™ 3.0 PK Suture Anchor with Needles: Yes | 70
  RAPTORMITE™ 3.0 PK Suture Anchor with Needles: No | 1
  FOOTPRINT™ ULTRA PK SL SUTURE ANCHOR: number analyzed (Participants) | 57
  FOOTPRINT™ ULTRA PK SL SUTURE ANCHOR: Yes | 57
  FOOTPRINT™ ULTRA PK SL SUTURE ANCHOR: No | 0

2. Secondary Outcome: Number of Participants With Clinical Success of the Study Devices in the Extremity Over a Time Period of 12 Months After Intervention
Description: Clinical success was defined as extremity repairs without signs of device failure and/or re-intervention as assessed by the surgeon. Specifically, clinical success was considered "Yes" based on the following 3 main criteria:
  * no inflammatory or allergic response
  * no device-related adverse event (AE)
  * no device deficiencies (DDs) leading to revision surgery (reintervention) on the index extremity
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Polyetheretherketone (PEEK) Extremity Suture Anchors
Number analyzed (Participants) | 23
Participants
  DYNOMITE™ 2.0 PK Suture Anchor With Needles: number analyzed (Participants) | 2
  DYNOMITE™ 2.0 PK Suture Anchor With Needles: Yes | 2
  DYNOMITE™ 2.0 PK Suture Anchor With Needles: No | 0
  RAPTORMITE™ 3.0 Suture Anchor With Needles: number analyzed (Participants) | 8
  RAPTORMITE™ 3.0 Suture Anchor With Needles: Yes | 8
  RAPTORMITE™ 3.0 Suture Anchor With Needles: No | 0
  FOOTPRINT™ Ultra PK SL Suture Anchor: number analyzed (Participants) | 16
  FOOTPRINT™ Ultra PK SL Suture Anchor: Yes | 16
  FOOTPRINT™ Ultra PK SL Suture Anchor: No | 0

3. Other Pre Specified Outcome: Visual Analog Scale (VAS) - Pain
Description: The VAS pain score is presented on a scale ranging from 0 to 10. A score of 0 represents no pain and a score of 10 indicates extreme/unbearable pain. The VAS rating was recorded retrospectively, per standard of care at 6 and 12 months post-surgery.
Time Frame: 6 and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Polyetheretherketone (PEEK) Extremity Suture Anchors
Number analyzed (Participants) | 48
score on a scale
  DYNOMITE™ 2.0 PK Suture Anchor With Needles: 6 months: number analyzed (Participants) | 1
  DYNOMITE™ 2.0 PK Suture Anchor With Needles: 6 months | 2 (NA) — Standard deviation not calculated whenever there was only 1 participant's data available
  DYNOMITE™ 2.0 PK Suture Anchor With Needles: 12 months: number analyzed (Participants) | 0
  RAPTORMITE™ 3.0 Suture Anchor With Needles: 6 months: number analyzed (Participants) | 13
  RAPTORMITE™ 3.0 Suture Anchor With Needles: 6 months | 1.8 (2.2)
  RAPTORMITE™ 3.0 Suture Anchor With Needles: 12 months: number analyzed (Participants) | 3
  RAPTORMITE™ 3.0 Suture Anchor With Needles: 12 months | 3.7 (4.0)
  FOOTPRINT™ Ultra PK SL Suture Anchor: 6 months: number analyzed (Participants) | 37
  FOOTPRINT™ Ultra PK SL Suture Anchor: 6 months | 2.6 (2.5)
  FOOTPRINT™ Ultra PK SL Suture Anchor: 12 months: number analyzed (Participants) | 12
  FOOTPRINT™ Ultra PK SL Suture Anchor: 12 months | 2 (2.8)

4. Other Pre Specified Outcome: Count of Participants With Range of Motion (ROM) Full Functional Arc
Description: Range of motion defined as the participant having a full functional arc "Yes" or "No" at 6 month and 12 month post-operative visits.
Time Frame: 6 and 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Polyetheretherketone (PEEK) Extremity Suture Anchors
Number analyzed (Participants) | 98
Participants
  DYNOMITE™ 2.0 PK Suture Anchor With Needles: 6 months: number analyzed (Participants) | 6
  DYNOMITE™ 2.0 PK Suture Anchor With Needles: 6 months: Has full functional arc: Yes | 3
  DYNOMITE™ 2.0 PK Suture Anchor With Needles: 6 months: Has full functional arc: No | 2
  DYNOMITE™ 2.0 PK Suture Anchor With Needles: 6 months: Has full functional arc: Unknown | 1
  DYNOMITE™ 2.0 PK Suture Anchor With Needles: 12 months: number analyzed (Participants) | 0
  RAPTORMITE™ 3.0 Suture Anchor With Needles: 6 months: number analyzed (Participants) | 55
  RAPTORMITE™ 3.0 Suture Anchor With Needles: 6 months: Has full functional arc: Yes | 21
  RAPTORMITE™ 3.0 Suture Anchor With Needles: 6 months: Has full functional arc: No | 5
  RAPTORMITE™ 3.0 Suture Anchor With Needles: 6 months: Has full functional arc: Unknown | 29
  RAPTORMITE™ 3.0 Suture Anchor With Needles: 12 months: number analyzed (Participants) | 6
  RAPTORMITE™ 3.0 Suture Anchor With Needles: 12 months: Has full functional arc: Yes | 1
  RAPTORMITE™ 3.0 Suture Anchor With Needles: 12 months: Has full functional arc: No | 2
  RAPTORMITE™ 3.0 Suture Anchor With Needles: 12 months: Has full functional arc: Unknown | 3
  FOOTPRINT™ Ultra PK SL Suture Anchor: 6 months: number analyzed (Participants) | 42
  FOOTPRINT™ Ultra PK SL Suture Anchor: 6 months: Has full functional arc: Yes | 34
  FOOTPRINT™ Ultra PK SL Suture Anchor: 6 months: Has full functional arc: No | 8
  FOOTPRINT™ Ultra PK SL Suture Anchor: 6 months: Has full functional arc: Unknown | 0
  FOOTPRINT™ Ultra PK SL Suture Anchor: 12 months: number analyzed (Participants) | 12
  FOOTPRINT™ Ultra PK SL Suture Anchor: 12 months: Has full functional arc: Yes | 11
  FOOTPRINT™ Ultra PK SL Suture Anchor: 12 months: Has full functional arc: No | 1
  FOOTPRINT™ Ultra PK SL Suture Anchor: 12 months: Has full functional arc: Unknown | 0

ADVERSE EVENTS:
Time Frame: Surgery to End of Study (EOS) visit, approximately 12 months
Description: AE reporting was collected retrospectively from the information available in the participant's medical records. A total of 140 participants were enrolled in the study. However, there were 2 participants with multiple devices implanted. Participant Suture Anchor data was analyzed independently based on the device implanted (i.e., participants implanted with multiple devices were analyzed individually based on unique suture anchor).
Groups:
- DYNOMITE™ 2.0 PK Suture Anchor With Needles: Participants who have received DYNOMITE™ 2.0 PK Suture Anchor with Needles
- RAPTORMITE™ 3.0 Suture Anchor With Needles: Participants who have received RAPTORMITE™ 3.0 Suture Anchor with Needles
- FOOTPRINT™ Ultra PK SL Suture Anchor: Participants who have received FOOTPRINT™ Ultra PK SL Suture Anchor
Arm/Group | DYNOMITE™ 2.0 PK Suture Anchor With Needles | RAPTORMITE™ 3.0 Suture Anchor With Needles | FOOTPRINT™ Ultra PK SL Suture Anchor
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/71 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/17 | 2/71 | 2/57
Other Adverse Events (participants affected / at risk) | 5/17 | 0/71 | 2/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DYNOMITE™ 2.0 PK Suture Anchor With Needles (N=17) | RAPTORMITE™ 3.0 Suture Anchor With Needles (N=71) | FOOTPRINT™ Ultra PK SL Suture Anchor (N=57)
SURAL NERVE DAMAGE AND MONONEUROPATHY/PAIN SYNDROME FROM POPLITEAL ANESTHETIC BLOCK. (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to device
HOSPITALIZATION FOR UTI, ACUTE RENAL FAILURE, SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) — Unrelated to device
COMPLEX REGIONAL PAIN SYNDROME (General disorders) | 0 (0) | 1 (1) | 0 (0) — Definitely related to device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DYNOMITE™ 2.0 PK Suture Anchor With Needles (N=17) | RAPTORMITE™ 3.0 Suture Anchor With Needles (N=71) | FOOTPRINT™ Ultra PK SL Suture Anchor (N=57)
LEFT ACHILLES CHRONIC PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to device
DEHISCENCE WOUND (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to device
PAIN OVER LATERAL ASPECT OF LEFT ANKLE (ONGOING AT 6 MONTHS). (General disorders) | 1 (1) | 0 (0) | 0 (0) — Unlikely related to device
PAIN OVER LATERAL ASPECT OF LEFT ANKLE AT 6 MONTHS (General disorders) | 1 (1) | 0 (0) | 0 (0) — Possibly related to device
SUPERFICIAL YEAST INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Unlikely related to device
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — Unrelated to device
FALL DOWN ON LEFT HEEL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Unrelated to device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT03782298/Prot_SAP_000.pdf